CLINICAL TRIAL: NCT06038214
Title: The Effect of Core Exercises on Pelvic Dysfunction, Sexual Dysfunction, Pain, Sleep Quality and Quality of Life in Women With Fibromyalgia
Status: Completed | Type: Observational
Sponsor: Inonu University (Other)
Collaborators: Burcu Talu (Unknown)
Responsible Party: Principal Investigator, Naciye Dilruba Tektas Gulbil, msc physiotherapist, Inonu University
Other Study IDs: 2022/3421
Record Dates: First submitted 2022-09-05; First posted 2023-09-14 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2024-03

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Exercise

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (2):
- core exercises grup: Core Exercise Group Exercises The exercise program was planned as warm-up, core exercises and cool-down periods, 2 days a week, 30 minutes a day and 8 weeks.
  In the warm-up and cool-down program, each exercise was planned as 3 sets of 10 seconds.
  The first 2 weeks of exercises were planned as 6 repetitions, the next 2 weeks the exercises 10 repetitions and the last 4 weeks the exercises were planned as 12 repetitions.
  Interventions: Other: core exercises
- home exercises grup: At the beginning of the study, it is planned to give a home exercise program for 30 minutes, 2 days a week for 8 weeks, with information and teaching home exercises at the beginning of the study. The content of the home exercise program will be therapeutic exercises, stretching and relaxation exercises.
  Evaluations will be evaluated for each group at the same time of the day before the exercise program starts and 1 day after the last session after completing 2 sessions a week for 8 weeks.
  Interventions: Other: home exercises

INTERVENTIONS:
Other: core exercises — 1.5 minutes walking 2. Stretching exercise
  * hallowing in supine and side lying position
  * Bracing in supine and side lying position
  * Bracing on the prone and forearms
  * Bracing in the crawling position
  * Bracing in laptop, half-lap and standing position
  * Heel slide exercise
  * Bridge building exercise
  * Unilateral limb flexion exercise in crawling position
  * Reciprocal heel slide exercise in supine position
  * Bilateral lower extremity lifting exercise
  * Unilateral lower extremity flexion in bridging position
  * Side bridging exercise with knees extended
  * Unilateral lower extremity extension in crawling position
  * Contralateral lower and upper extremity lift in the crawling position
  * Straight and oblique trunk flexion
  * Straight and oblique trunk flexion with hip and knee flexed to 90°
  * bracing on the ball
  * squat
  * bracing while walking
  Other Names: exercises
  Groups: core exercises grup
Other: home exercises — Right and left rotation of the head
  * lateral flexion of the head
  * Flexion and extension of the head
  * Stretching the neck extensors
  * pectoral stretch
  * Stretching the hip extensors
  * Hamstrig stretching
  * Stretching the lumbar extensors
  * Abdominal strengthening
  * bridging
  * Hip abduction strengthening
  * hip extension strengthening
  * Upper extremity resistant flexion
  * Upper extremity resistant abduction
  * Upper extremity relaxation exercise
  * Capsule stretching
  * Stretching the hip flexors
  * Stretching the lower extremity adductors
  * relaxation exercise
  Groups: home exercises grup

SUMMARY:
In fibromyalgia patients, exercise is needed to reduce symptoms and to prevent muscle weakness with fatigue and pain. Core exercise retrains and strengthens deep postural spinal muscles such as the multifidus and transverse abdominis by promoting neuromuscular control, maintaining the dynamic stability of the spine and thus reducing pain. By performing core exercises, the pelvic floor, which forms the lower base of the core, is strengthened.

Objective: It was planned to investigate the effects of core exercises on pelvic floor dysfunction, sexual dysfunction, pain, sleep quality and quality of life in women with fibromyalgia.

Materials and Methods: It was designed as randomized control. Sexually active women with fibromyalgia syndrome between the ages of 18-65 will be included in the study. After the patients are selected from the relevant stage with the improbable random sampling method, the patients who accept to participate in the study and meet the inclusion criteria will be assigned to one of the groups in which the core exercise or home program is applied. Evaluations will be evaluated for each group before starting the exercise program and 1 day after the last session, following the completion of 2 sessions per week for 8 weeks. Pain Visual Analog Scale; fibromyalgia impact level Revised Fibromyalgia Impact Questionnaire (FIQR); pelvic floor dysfunction Pelvic Floor Impact Questionnaire (PFIQ); sexual dysfunction Female Sexual Function Scale; sleep quality: Pittsburgh Sleep Quality Index; short quality of life It is planned to be evaluated with Form-36(SF-36). Conclusion: The effects of core exercises on pelvic floor dysfunction, sexual dysfunction, pain, sleep quality and quality of life will be evaluated and interpreted by comparing the evaluations before and after treatment and between groups.

DETAILED DESCRIPTION:
Fibromyalgia (FM) is a non-articular, chronic rheumatic disease of unknown etiology, characterized by widespread musculoskeletal pain, sleep disturbance, mood changes, fatigue, and the presence of multiple tender points. Diagnostic criteria were defined by the American Rheumatism Association (ARA) in 1990. To diagnose FM, there should be widespread pain and tenderness at 11 or more of 18 specific points (1).

Although the etiopathogenesis of FM is still unknown, triggering factors such as physical trauma, surgical intervention, infections, acute or chronic emotional stress may play a role (2). Various findings such as muscular symptoms accompanying chronic pain, cognitive complaints, depression, insomnia and fatigue have been described in patients with FM (2). chronic pain seen in FM; It creates physical and emotional stress such as sleep, fatigue and cognitive symptoms. In addition, unwillingness to move or fear of movement may develop in individuals due to chronic pain (2).

Various psychopathological disorders have been reported in FM. It is estimated that 1/3 of his patients have minor depression or anxiety and anxiety state disorder. However, it is unknown whether anxiety and depression in FM cause chronic pain or contribute to the severity of symptoms (1). Despite various complaints of patients with fibromyalgia, the absence of a significant disorder in physical examination and laboratory tests suggests that the symptoms may be of psychological origin (2). Since the etiology of fibromyalgia syndrome is unknown, pharmacological and non-pharmacological treatment methods should be used in patient-specific combinations according to the prominent symptoms and their severity (2).

Sexuality is an important part of life and is associated with the well-being of the individual. Sexuality covers many issues, starting with the self-image of the person and the relationship with his partner (3). Sexual dysfunction is defined as the satisfaction of not participating in sexual acts (3). The development of sexual dysfunction in women with fibromyalgia is thought to be associated with many factors such as symptoms, pain, anxiety, depression, and drug therapy (3).

Few studies have been done on the sexuality of women with fibromyalgia (4), and studies have found a relationship between fibromyalgia and sexual dysfunction (4) In addition, considering that women with fibromyalgia have an increase in pain, fatigue, and decrease in muscle strength (5), Fusco et al. concluded that women with fibromyalgia exhibited weaker pelvic floor muscles and also more frequent lower urinary tract symptoms compared to the healthy control group (5). For this reason, a relationship between pelvic floor involvement and impaired sexual function in women with fibromyalgia is considered (5).

It is reported that sleep quality is deteriorated by almost 80% of patients with fibromyalgia (6). Epidemiological studies show that poor sleep quality is a risk factor for fibromyalgia. Poor sleep is associated with symptom severity in patients with fibromyalgia (6). It has been shown that improving sleep quality in exercise approaches as well as pharmacological treatments can reduce pain in patients with fibromyalgia (6,7).

When looking at the quality of life, studies comparing the quality of life in FM patients with healthy individuals of the same age show that FM has a negative effect, as symptoms affect daily routine and physical activities, causing patients to enter a vicious circle(8). Because fibromyalgia has a negative effect on fatigue, pain, anxiety, sleep disturbance symptoms, and poor quality of life, the American Pain Society and the Association of Scientific Medical Societies in Germany have recommended physical exercise, hydrotherapy, massage, yoga and various treatment strategies besides medication use. It is recommended in methods such as acupuncture (9).

The term core is used for the trunk or more specifically the lumbopelvic region of the body. Stabilization of the lumbopelvic region is very important for upper and lower extremity movements, supporting loads, protecting nerve roots and spinal cord. (10,11). core; It can be thought of as a box formed by the abdominals in the front, the paraspinals and gluteals in the back, the diaphragmatic roof above, and the pelvic floor muscles at the bottom. When the stabilization system works effectively, optimal control and efficiency of the movement, proper distribution of the force, adequate absorption of the ground effect force and protection of the joints in the kinetic chain are ensured. (12,13). The stabilization system consists of 3 sub-systems as neural, passive and active systems and are functionally interconnected (11). The neural system receives stimuli from the muscle spindle, Golgi tendon organ and spinal ligaments, adjusts the muscle strength, and determines the spinal stability requirements. Stability can change abruptly depending on the external loads that the body can carry along with postural adjustments. The neural system has to work synchronously with other systems in order to perform the desired movement and to provide sufficient stability (11). The passive system consists of spinal ligaments and facet joints and allows limited loading of the lumbar vertebrae. For this reason, an active system is needed to load and support body mass in resistant exercise-dynamic activities (11). The active system consists of muscles and tendons. The active musculature, on the other hand, has been divided into two as "global" and "local" according to their roles in core stabilization (11). The global group consists of large superficial muscles. The muscles in the global musculature are the erector spina, external oblique, and rectus abdominis (10). The local group is; It consists of deep and small muscle groups. The local musculature consists of transversus abdominus, multifidi, internal oblique, deep transversospinalis and pelvic floor muscles (10). For the continuity of spinal function, the simultaneous function of the global and local groups is required (13). Core muscles consist of 2 types of muscle fiber structures that contract slowly and quickly. Slow-twitch fibers are mainly located in the local system known as the deep layer, providing intersegmental movement control and posture changes. Fast-twitch fibers are found in the superficial layer, that is, in the global musculature. These muscles are fibers with large torque capability focused on speed, power, and greater range of motion (10-13). Pelvic floor muscles form the base of the core muscles. The pelvic floor not only plays an important role in muscle activation for lumbar stabilization, but also forms the basis of the abdominal cavity. Pelvic floor muscles; During work that increases intra-abdominal pressure, it should contract in order to maintain continence and contribute to the increase in pressure (14). It has been reported that the contraction of the pelvic floor muscles can be strengthened by the activation of the trunk stabilizing muscles. Therefore, trunk stabilization exercises are thought to be an option to increase the effectiveness of pelvic floor muscle exercises (15).

Pelvic floor dysfunction is defined as the abnormal function of the pelvic floor and includes conditions that may have significant adverse effects on a woman's quality of life, such as urinary incontinence (stress, urge, and mixed), fecal incontinence, pelvic organ prolapse, and sexual dysfunction (16).

Core exercise is recommended in the rehabilitation of chronic pain (17). Few studies on the management of pain in fibromyalgia have focused on core exercise (18). The main purpose of core exercise is to promote neuromuscular control and retrain and strengthen the deep postural spinal muscles such as the multifidus and transversus abdominis, maintain the dynamic stability of the spine and thus reduce pain (19,20). Core exercise alone reduced pain and depression and improved health status, quality of life and sleep quality in women with FM(19-22).

Core exercise focuses on activating the deep local musculature, regulating overactivity of surface muscles, and restoring normal synergistic function between local and global musculature, thereby reducing pain and improving function (19,21). Although the positive effects of core exercise on chronic pain such as low back pain are well known (21), the number of studies focusing on core exercise in axial pain, which is common in FM, is insufficient. Only one study in the literature focused on investigating the effects of specific core exercise on FM (18). Martinez-Rodriguez et al. (18) recently found that core exercise plus lacto-vegetarian diet contributed to the reduction of pain and improvement of body composition in FM. The current study reveals that core exercise alone is effective in reducing pain and depression and improving health status, quality of life and sleep quality in FM.

When we look at the literature, many studies have revealed that the symptoms of fibromyalgia syndrome such as fatigue, depression, pain and sleep disturbance are also associated with sexual dysfunction by affecting the pelvic floor (8). In line with this information, our aim is to examine the effects of core exercises on pelvic floor dysfunction, sexual dysfunction, pain, sleep quality and quality of life in women with fibromyalgia.

5.1. Type of study: Experimental randomized controlled trial 5.2. Place and time of the research: İnönü University Turgut Özal Medical Center Department of Rheumatology 20.06.2022-20.12.2023 5.3. The universe and sample of the research: The population of the study, which was planned as a randomized controlled study, consists of sexually active women with fibromyalgia syndrome by the relevant specialist physician of İnönü University Turgut Özal Medical Center Rheumatology Department. For the study, which is planned to be carried out between 20.06.2022 and 20.12.2023, after the patients are selected from the relevant stage with the improbable random sampling method, the patients who accept to participate in the study and meet the inclusion criteria will be assigned to one of the groups in which core exercise or home program is applied.

Inclusion criteria for the study:

Be between the ages of 18 and 60 with a previous diagnosis of fibromyalgia Symptoms last longer than 3 months Being sedentary (not doing physical activity at least 3 days a week in the last 3 months) being sexually active To voluntarily accept participation in an exercise program 2 days a week for 8 weeks,

Exclusion criteria from the study:

Using psychotropic medication in the last 1 month Known central or peripheral nervous system disease, progressive neurological damage, Presence of any cardiovascular pathology, Presence of uncontrolled hypertension, Presence of any musculoskeletal system disease other than fibromyalgia, Pregnancy, Presence of cognitive problems that will affect cooperation

Exclusion criteria:

Volunteer's request to leave Failure to continue training sessions

5.4. Study material: Evaluations will be evaluated for each group before starting the exercise program and 1 day after the last session, following the completion of 2 sessions per week for 8 weeks. Pain Visual Analog Scale; fibromyalgia impact level Revised Fibromyalgia Impact Questionnaire (FIQR); pelvic floor dysfunction Pelvic Floor Impact Questionnaire (PFIQ Pelvic Floor Impact Questionnaire); sexual dysfunction Female Sexual Function Scale; sleep quality: Pittsburgh Sleep Quality Index; It is planned to evaluate the quality of life with Short Form-36 (SF-36).

5.5. Data collection tools: Data Collection Inonu University Turgut Özal Medical Center Rheumatology Department diagnosed with fibromyalgia by the relevant specialist, sexually active women between the ages of 18-65 will be included in the study. Individuals will be evaluated for compliance with the study content before the preliminary evaluation. After eligibility is determined, individuals will be randomly assigned to groups. In the randomization of the groups, the assignment will be made to the groups with the randomizer program using the computer. Evaluations will be evaluated for each group at the same time of the day before the exercise program starts and 1 day after the last session after completing 2 sessions a week for 8 weeks.

Evaluation form : Sociodemographic data of individuals will be questioned with an evaluation form. Evaluation form; patient's name-surname, age, gender, height, weight, marital status and duration of marriage, age at diagnosis and education level.

Pain: Regional neck and back pain at rest and during activity will be evaluated with the help of the Visual Analogue Scale (VAS). The VAS is a 10 cm scale that rates 0 points as "no pain" and 10 points as "worst pain imaginable".

Fibromyalgia Impact Level : Revised Fibromyalgia Impact Questionnaire (FIQR) will be used. This scale; physically It measures 10 different features: function, well-being, not being able to go to work, difficulty at work, pain, fatigue, morning fatigue, stiffness, anxiety and depression. With the exception of the well-being trait, low scores indicate recovery or less affliction. FEA is filled by the patient. The maximum possible score of each sub-title is 10. Thus the total maximum score is 100. The average FM patient scores 50, while more severely affected FM patients usually score above 70. Permission to use the survey has been obtained.

Pelvic floor assessment: Pelvic Floor Impact Questionnaire (PFIQ Pelvic Floor Impact Questionnaire) will be used for measurement. The PFIQ is a pelvic floor quality of life questionnaire used to evaluate the effects of bowel, bladder, and/or pelvic symptoms on an individual's activities of daily living, social relationships, and emotions. Each item consists of 4 options (Never, Rarely, Moderately, Quite often) and is scored between 0 and 3. The PFIQ scale also consists of 3 sub-dimensions. POPIQ-7 (Pelvic organ prolapse impact questionnaire): In this sub-dimension consisting of 7 questions, it is questioned how the pelvic organ prolapse affects the patient during travel, social activity and physical activity and the effect of this situation on emotional health. CRAIQ-7 (Colo-rectal-anal impact questionnaire): In this sub-dimension consisting of 7 questions, it is questioned how intestinal complaints affect the patient during travel, social activity and physical activity and the effect of this situation on emotional health. The mean scores of the items in each sub-dimension are calculated and these scores are multiplied by (100/3) and PFIQ subscale scores ranging from 0-100 are calculated. Then, the 3 subscale scores are summed to find the PFIQ total score, which ranges from 0-300. A higher score indicates worse health. Permission to use the survey has been obtained.

Sexual Dysfunction: It will be measured with the Female Sexual Dysfunction Scale. The scale consists of 19 questions. Each The question has six options to answer, and each item is scored from zero to five. In the structure of the scale; There are six sub-dimensions: desire, arousal, lubrication, orgasm, satisfaction and pain. The person gets a score between 4 and 95 from the scale. Permission to use the survey has been obtained.

Sleep Quality: Pittsburgh It will be measured by the Sleep Quality Index. Defining good and bad sleep and assesses sleep quality. It consists of a total of 24 questions, 19 of which are self-evaluation and 5 of which are answered by the spouse or roommate of the person. The questions are collected in 7 subscales. These are: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleeping pills, and daytime dysfunction. Each subscale is scored between 0-3 points. The total score is between 0-21. Questions asked to an individual's spouse or roommate are not included in the calculation. Permission to use the survey has been obtained.

Quality of life: The Short Form-36 (SF-36) scale will be used. Assessing the SF-36 quality of life developed for the purpose. A validity and reliability study was conducted in Turkey. SF-36 is used to compare general and specific populations, to demonstrate the health benefits of different treatments, and to monitor patients. The last 4 weeks are taken into account in the evaluation of SF-36, which consists of a total of 36 items. It is stated that due to the release of SF-36 v2.0, the use of v1.0 does not require permission.

5.6. Variables of the research While the dependent variables of our study were pelvic floor dysfunction, sexual dysfunction, pain, sleep quality and quality of life, the independent variables were age, gender, height, weight, marital status and duration of marriage, age at diagnosis, and education level.

5.7. research plan The population of the study, which was planned as a randomized controlled study, consists of sexually active women with fibromyalgia syndrome by the specialist physician of the Inonu University Turgut Özal Medical Center Rheumatology Department. For the study, which is planned to be carried out between 20.06.2022 and 20.12.2023, after the patients are selected from the relevant stage with the improbable random sampling method, the patients who accept to participate in the study and meet the inclusion criteria will be assigned to one of the groups in which core exercise or home program is applied.

Treatment protocol:

The individuals included in the study will be divided into 2 groups.

* Group (experiment): Individuals in this group are planned to be included in the core exercise program.
* Group (control): It is planned to receive a follow-up home program and information.

The core exercise group will be included in the exercise program under the supervision of a physiotherapist, with 30 minutes each session, 2 days a week for 8 weeks. 30-minute exercise sessions are planned as 5 minutes of warm-up, 20-minutes of core exercises and 5 minutes of cool-down.

ELIGIBILITY:
Inclusion Criteria

* Be between the ages of 18 and 60 with a previous diagnosis of fibromyalgia
* Symptoms last longer than 3 months
* Being sedentary (not doing physical activity at least 3 days a week in the last 3 months)
* being sexually active
* To voluntarily accept participation in an exercise program 2 days a week for 8 weeks,

Exclusion criteria from the study

* Using psychotropic medication in the last 1 month
* Known central or peripheral nervous system disease, progressive neurological damage
* Presence of any cardiovascular pathology
* Presence of uncontrolled hypertension
* Presence of any musculoskeletal system disease other than fibromyalgia
* Pregnancy
* Presence of cognitive problems that will affect cooperation

Exclusion criteria:

* Volunteer's request to leave
* Failure to continue training sessions

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: fibromiyalgia
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-05-20 (Actual)

PRIMARY OUTCOMES:
Pelvic Floor Impact Questionnaire (PFIQ ) | 8 weeks
  Pelvic floor assessment: Pelvic Floor Impact Questionnaire (PFIQ) Pelvic Floor Impact Questionnaire) will be used for measurement. PFIQ is a pelvic floor quality of life questionnaire used to assess the effects of bowel, bladder, and/or pelvic symptoms on an individual's activities of daily living, social relationships, and emotions.
Female Sexual Dysfunction Scale | 8 weeks
  Sexual Dysfunction: Will be measured by the Female Sexual Dysfunction Scale. The scale consists of 19 questions. Each question has six options that need to be answered, and each item is scored from zero to five. In the structure of the scale; There are six sub-dimensions: desire, arousal, lubrication, orgasm, satisfaction, and pain. The person scores between 4 and 95 on the scale. Permission has been obtained to use the survey.
Visual Analog Scale (VAS) | 8 weeks
  Pain: Regional neck and back pain during rest and activity will be evaluated with the help of Visual Analog Scale (VAS). The VAS is a 10cm scale that evaluates 0 points as "no pain" and 10 points as "the worst pain imaginable".
Pittsburgh Sleep Quality Index | 8 weeks
  Sleep Quality: Will be measured by the Pittsburgh Sleep Quality Index. Identification of good and bad sleep and assessment of sleep quality. It consists of a total of 24 questions, 19 of which are self-assessment and 5 of which are answered by the person's spouse or roommate. The questions are collected in 7 sub-scales. These; subjective sleep quality, sleep delay, sleep duration, habitual sleep activity, sleep disturbance, sleep medication use and daytime dysfunction. Each subscale is scored between 0-3 points. The total score is from 0-21. Questions asked to an individual's spouse or roommate are not included in the calculation. Permission has been obtained to use the survey
Short Form-36 (SF-36) | 8 weeks
  Quality of life: Short Form-36 (SF-36) scale will be used. Evaluation of the quality of life of SF-36 developed for this purpose. Validity and reliability studies were conducted in Turkey. SF-36 is used to compare general and specific populations, demonstrate the health benefits of different treatments, and monitor patients. In the evaluation of KF-36, which consists of a total of 36 items, the last 4 weeks are taken into account. Due to the release of the SF-36 v2.0, the use of v1.0 does not require permission.

CONTACTS AND LOCATIONS:
Locations (1):
- Inonu Unıversity, Malatya, Malatya, Turkey (Türkiye)